CLINICAL TRIAL: NCT03442595
Title: Expanded MedStar Diabetes Pathway Ongoing Chart Review Protocol
Brief Title: MedStar Diabetes Pathway Chart Reviews
Acronym: MedstarBC2
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Michelle Magee, Director, MedStar Diabetes Institute, Medstar Health Research Institute
Other Study IDs: 2016-143
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: patients with uncontrolled type 2 diabetes mellitus that participate in the MedStar Diabetes Pathway
  Interventions: Other: Intensive diabetes education and medication management
- Matched controls: patients with uncontrolled type 2 diabetes that match the cases on 5 criteria and received standard of care diabetes management with a MedStar provider

INTERVENTIONS:
Other: Intensive diabetes education and medication management — Patients receive intensive knowledge based diabetes education and algorithm driven medication management over a period of 12 weeks.
  Groups: Cases

SUMMARY:
The MedStar Diabetes Pathway (MDP) is transitioning into a clinical program offered at various MedStar sites. The MDP clinical team is reviewing the data collected during the pilot to improve the program and adapt it to various clinical settings in order to better serve the target patient population. It is imperative to continue reviewing patient clinical outcomes as the program expands in order to insure continuous quality improvement of the program. This will be achieved through chart reviews of patients receiving diabetes care via the MDP and comparison with patients received diabetes standard of care through their primary care physician.

DETAILED DESCRIPTION:
The MedStar Diabetes Pathway (MDP) early pilot program has generated evidence that an innovative technology-enabled "Boot Camp" approach to the delivery of diabetes survival skills education and medication management has a significant impact on glycemic control and healthcare utilization measures. The MDP is a 12 week Diabetes "Boot Camp" technology-enabled intervention which will offer learner-centered survival skills self-management education (DSSE) and algorithm-driven diabetes medications (DM) titration by Endocrinologist-supervised Certified Diabetes Educators (CDE), NPs and PharmDs. The program has been offered at 5 MedStar Medical Group (MMG) Primary Care Practices from November 2014 to February 2016 to high risk adults with uncontrolled type 2 diabetes who have a hemoglobin A1C (A1C) level -a marker of average blood glucose (BG) levels in the 2-3 months prior to the time the test is done- which is at or above 9% - considered to be poor control, and 1 or more additional risk factors for poor health outcomes. The program has been well received by MedStar Primary Care Providers and their diabetes patients. Patients that participated in the MDP achieved significantly higher A1C reduction and decreased risk risk for acute care utilization then matched controls that received standard of care. The pilot evidence demonstrated a significant impact on glycemic control and healthcare utilization measures as the result of a concise, focused DM education and medication management intervention. Building on the success of the MDP Phase 1.0 pilot, the next steps in expanding the program will be as follows:

* Transition of the Pathway from early feasibility pilot to the next phase as an expanded pilot program integrated within the MedStar Health System care delivery network and built upon a sustainable infrastructure across early adopter MMG practice sites.
* Expand recruitment to include high risk patients with uncontrolled type 2 diabetes, including those with a new diagnosis and A1C >9%, who have MedStar Emergency Department and/or Inpatient encounters
* Spread to additional targeted MedStar Primary Care Practices and/or to MedStar Managed Care Plan participants.

Chart reviews and data collection during the expansion phase will be essential to guide the process and allow rapid cycle adjustments to maximize the impact of the program and utilization of resources for the benefit of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes, A1C equal or higher than 9%, active patient of medstar health provider, english speaking, willing and able to participate in the program

Exclusion Criteria:

* A1C less than 9%, severe illness that precludes participation such severe congestive heart failure or COPD, advanced kidney disease, recent acute illness such as heart attack or stroke in the past 30 days, active cancer, severe mental illness, high dose steroid, other types of diabetes, pregnant or lactating.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with uncontrolled type 2 diabetes that meet inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Magee, MD, Principal Investigator — Medstar Health Research Institute

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Matched Controls
Started | 460 | 366
Completed | 366 | 366
Not Completed | 94 | 0
Not completed — Lost to Follow-up | 94 | 0

BASELINE CHARACTERISTICS:
Population: A total of 460 patients started the diabetes boot camp (cases) during the study period, but only 366 completed it and were included in the results analysis.
Groups:
- Cases: Adult patients with uncontrolled type 2 diabetes mellitus and A1C>/= 9% that participate in the MedStar Diabetes Pathway
  Intensive diabetes education and medication management: Patients receive intensive knowledge based diabetes education and algorithm driven medication management over a period of 12 weeks.
- Concurrent Matched Controls: Adult patients with uncontrolled type 2 diabetes and A1C>/=9% that propensity match the cases on 5 criteria and received standard of care diabetes management with a MedStar provider
- Total: Total of all reporting groups
Arm/Group | Cases | Concurrent Matched Controls | Total
Number analyzed (Participants) | 366 | 366 | 732
Age, Categorical [Count of Participants; unit: Participants] — Population: 460 patients were enrolled but only the 366 that completed the boot camp were included in the analysis
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 293 | 293 | 586
    >=65 years | 73 | 73 | 146
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 460 patients were enrolled but only the 366 patients that completed the boot camp were included in the analysis
  Participants
    Female | 225 | 233 | 458
    Male | 141 | 133 | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 460 patients were enrolled but only the 366 that completed the boot camp were included in the analysis
  Participants
    Hispanic or Latino | 4 | 3 | 7
    Not Hispanic or Latino | 362 | 363 | 725
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 460 patients were enrolled but only the 366 patients that completed the boot camp were included in the analysis
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 4 | 4 | 8
    Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
    Black or African American | 296 | 284 | 580
    White | 48 | 53 | 101
    More than one race | 5 | 5 | 10
    Unknown or Not Reported | 9 | 18 | 27
Region of Enrollment [Number; unit: participants] — Population: 460 were enrolled but only the 366 patients that completed the boot camp were included in the final analysis of results.
  participants
    United States | 366 | 366 | 732
Hemoglobin A1C >/=9% [Mean (Standard Deviation); unit: %] — Population: A total of 460 patients started the diabetes boot camp (cases) during the study period, but only 366 completed it and were included in the results analysis.
  % | 11.2 (1.7) | 11.3 (1.6) | 11.23 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in A1C
Description: Change in Hemoglobin A1C from baseline to 12-16 weeks for both cases and controls
Time Frame: 12-16 weeks
Population: Hemoglobin A1C was measured at baseline and at 3 months in both groups.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
% change | -3.06 (1.98) | -1.44 (2.11)
Statistical Analysis 1: Comparison: Cases vs Matched Controls; The study was powered to detect a difference of 0.5% in the change in A1C with SD = 2 with 80& at alopha = 0.;05 with a sample size of 128 in each group (paired t-test). The study reaches 100% power to detect this observed difference with an alpha level of 0.01; Test type: Other — test of difference in change of A1C between the two groups; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Risk for Emergency Room Visits at 30 Days From Baseline as Measured by Incidence Risk Ratio
Description: Comparison of risk of incurring an emergency room visits at 30 days from baseline for cases and controls. This was done by calculating and comparing the incidence risk ratio for an ER visit for each group and comparing them.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
ratio of risk incidences | 0.79 [0.42 to 1.47] | 0.39 [0.22 to 0.71]

3. Secondary Outcome: Risk for Hospitalizations at 30 Days From Baseline
Description: Comparison of risk for experiencing a hospital visit within 30 days from baseline in both group. This was done by calculating the incidence risk ratio for hospitalizations for cases and controls at 30 days from baseline and comparing them.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
ratio of risk incidences | 0.21 [0.07 to 0.60] | 1.14 [0.47 to 2.75]

4. Secondary Outcome: Risk for Composite of Emergency Room Visits and Hospitalizations at 30 Days From Baseline
Description: Comparison for risk of experiencing a visit to the emergency room and/or the hospital at 30 days from baseline. This was measured by calculating the Incidence risk ratio for acute care utilization at 30 days from baseline for both cases and controls and comparing them.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
ratio of risk incidences | 0.55 [0.34 to 0.90] | 0.53 [0.33 to 0.84]

5. Secondary Outcome: Risk for Emergency Room Visits at 90 Days From Baseline
Description: Comparison of the risk of experiencing an emergency room visit at 90 days from baseline in both groups. This was done by calculating the Incidence risk ratio for an emergency room visit at 90 days for both cases and controls and comparing them
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
ratio of risk incidences | 0.62 [0.42 to 0.92] | 0.66 [0.45 to 0.96]

6. Secondary Outcome: Risk for Hospitalizations at 90 Days From Baseline
Description: Comparison of the risk for experiencing a hospitalization within 90 days from baseline in both groups. This was done by calculating the Incidence Risk Ratio for hospitalizations for cases and controls within 90 days of baseline and comparing them.
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
ratio of risk incidences | 0.23 [0.11 to 0.50] | 1.58 [0.75 to 3.33]

7. Secondary Outcome: Composite of Risk for Hospitalizations and Emergency Room Visits Within 90 Days From Baseline
Description: Comparison of the risk for experiencing a hospitalization and/or emergency room visit within 90 days from baseline for both groups. This was done by calculating then comparing the incidence risk ratio for acute care utilization within 90 days from baseline for cases and controls.
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Cases | Matched Controls
Number analyzed (Participants) | 366 | 366
ratio of risk incidences | 0.49 [0.36 to 0.67] | 0.80 [0.58 to 1.10]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 90 days that patients were enrolled in the diabetes boot camp
Description: The definition of adverse events used was the same as from clinicaltrials.gov. Deaths and adverse events were not monitored/assessed for the matched controls as these patients were receiving diabetes standard of care and the matching was performed once the cases had completed the intervention.
Arm/Group | Cases
All-Cause Mortality (participants affected / at risk) | 0/460
Serious Adverse Events (participants affected / at risk) | 5/460
Other Adverse Events (participants affected / at risk) | 3/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cases (N=460)
worsening pre-existing heart failure (Cardiac disorders) | 1 (1) — Patient with preexisting class III/IV heart failure required hospitalization and LVAD placement. Was withdrawn from the boot cam due to extended hospital stay
Chest pain requiring hospitalization (Cardiac disorders) | 2 (2) — Patient with know history of CHF and CADA.
New diagnosis of breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — AE classified as unrelated to Boot Camp as patient had not been started on any new medications. Patient self-withdrew from the Boot Camp after receiving diagnosis and was lost to follow up.
Deep vein Thrombosis requiring intervention (Vascular disorders) | 1 (1) — Patient had a history of vascular problems
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cases (N=460)
Diabetic neuropathy (Musculoskeletal and connective tissue disorders) | 3 (3) — New diagnosis of diabetic neuropathy in patients with long standing type 2 DM

LIMITATIONS AND CAVEATS:
By design this was a real-world study and not a randomized controlled trial. The researchers chose a pragmatic study design over an RCT to see if the intervention was effective in real world situations under usual patient care conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03442595/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03442595/SAP_001.pdf